CLINICAL TRIAL: NCT00355355
Title: A Phase 3 Randomized Study to Evaluate Survival of Patients Treated With Talaporfin Sodium (LS11) and Interstitial Light Emitting Diodes (LED) as Compared to the Standard of Care Therapies in the Treatment of Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: A Phase 3 Study of Talaporfin Sodium and Interstitial Light Emitting Diodes Treating Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Light Sciences Oncology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSO-OL005
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Carcinoma, Hepatocellular; Liver Neoplasms
Keywords: Hepatocellular carcinoma; HCC; Liver Neoplasms; Talaporfin Sodium (LS11); Light emitting diodes (LEDs); Light activation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Talaporfin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Litx (Experimental): Drug: Talaporfin Sodium (1 mg/kg iv), Device: Interstitial Light Emitting Diodes (200 J/cm) 3 treatments within 6 months
  Interventions: Drug: Talaporfin sodium; Device: Interstitial Light Emitting Diodes; Procedure: Percutaneous placement of device in the liver
- Standard Care (Active Comparator): The standard of care could include any one of the following treatment options: Percutaneous Ethanol Injection (PEI), Transcatheter Arterial Chemoembolization (TACE), Radio Frequency Ablation (RFA), Cryotherapy, Systemic Chemotherapy, or other modalities that may be used at a particular institution.
  Interventions: Procedure: Standard Care

INTERVENTIONS:
Drug: Talaporfin sodium — LS11 (Talaporfin Sodium) slowly administered (3-5 min.) in a free flowing intravenous drip at a dose of 1 mg/kg.
  Arms: Litx
Device: Interstitial Light Emitting Diodes — 200 J/cm per Light Source at 20 mW/cm light energy
  Arms: Litx
Procedure: Percutaneous placement of device in the liver — Litx™ treatment group undergo CT or Ultrasound guided percutaneous placement of a single, two, three, or four Light Sources depending on their tumor characteristics. No more than 4 Light Sources will be used at a single treatment. The Light Source(s) may be used in a single lesion or in multiple lesions.
  Arms: Litx
Procedure: Standard Care — The standard of care could include any one of the following treatment options: Percutaneous Ethanol Injection (PEI), Transcatheter Arterial Chemoembolization (TACE), Radio Frequency Ablation (RFA), Cryotherapy, Systemic Chemotherapy, or other modalities that may be used at a particular institution.
  Arms: Standard Care

SUMMARY:
The purpose of the study is to assess the survival of patients treated with Litx™ versus standard of care therapies in the treatment of unresectable hepatocellular carcinoma (HCC), and to demonstrate the safety of Litx™ therapy.

Litx™ consists of a light-activated drug, talaporfin sodium (LS11, Light Sciences Oncology, Bellevue, Washington), and a light generating device, composed of light-emitting diodes (LEDs), that is energized by a power controller and percutaneously placed in the target tissue inside the body.

DETAILED DESCRIPTION:
Patients who provide Informed Consent and satisfy the Eligibility Criteria will be placed in an eligibility pool for randomization for either the Litx™ treatment arm or the standard of care arm.

A Patient assigned to the Litx™ treatment group may receive up to three Litx™ treatments. Regardless of which group the patient is assigned the treatment planning should anticipate ablation of all lesions with three Litx™ treatments using up to 4 Light Sources per treatment (a single Light Source may kill 2 cm x 4 cm of tissue).

The Litx™ treatment group undergo CT or Ultrasound guided percutaneous placement of a single, two, three, or four Light Sources depending on their tumor characteristics. No more than 4 Light Sources will be used at a single treatment. The Light Source(s) may be used in a single lesion or in multiple lesions. Following imaging confirmation of Light Source placement, patients will receive an intravenous dose of LS11 at 1 mg/kg. Fifteen minutes to one hour following completion of LS11 administration, delivery of 200 J/cm per Light Source at 20 mW/cm light energy will begin. The Light Source will then be manually removed and the patients will be observed for any complication after Light Source removal. Precautions for protection from external light exposure should be instituted beginning with the LS11 administration and maintained for up to two weeks.

Patients designated for the standard of care group, will receive current standard of care treatment recommended by the investigating physician. Should the elected treatment fail, a patient may switch to another standard of care treatment.

A patient designated for the Litx™ treatment group may receive up to two additional Litx™ treatments. A second and third treatment with Litx™ may be considered if any residual tumor or new tumor exists. The third treatment must take place within six months after the first treatment. A patient may switch to receiving standard of care after the third Litx™ treatment or as recommended by the investigator as necessary.

For either the Litx™ group or standard of care group once all treatment therapies have been exhausted the patient will be followed for survival. No protocol-directed office visits are required during this period and the patient may be followed by phone and/or e-mail at four week intervals. All patients will be monitored for survival from the time of randomization to the time of death from any cause or until at least 142 deaths have been observed, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of primary Hepatocellular Carcinoma (HCC), established by any one of the following criteria in a clinical setting suggestive of HCC: A. Two different imaging techniques with characteristics that suggest HCC; B. Combination of one imaging technique that suggests HCC and serum AFP level >400 ng/mL; C. Histological evidence of HCC
* ECOG Performance Status 0-2
* Life expectancy of at least 16 weeks
* Patients may have received previous antineoplastic therapy; at least 3 weeks must have elapsed since the completion of any prior therapy and the patient must have recovered from acute side effects.
* Understanding and ability to sign written informed consent
* 18 years of age or more
* Adequate hematologic, liver and renal functions as evidenced by the following: WBC >= 2,400/mm³ ; Platelet Count >= 75,000/µl ; Hemoglobin >= 9.4 gm/dL ; PT and PTT <= 1.5 Control ; SGOT, SGPT <= 5 × ULN ; Bilirubin <= 2.5 × ULN ; Alk Phos <= 3 × ULN ; Creatinine <= 2.5 mg/dL (SI: 221 mmol/L) ; Albumin >= 2 g/dL

Exclusion Criteria:

* Patients who are candidates for surgery with curative intent are not eligible
* Patients with 6 or more lesions are not eligible
* Patients with greater than 50% of parenchyma disease involvement are excluded
* Patients with Child-Pugh C cirrhosis are excluded
* Patients with diffuse HCC are excluded
* Patients with grade 3 ascites are excluded
* Evidence of major vessel invasion or extrahepatic disease is excluded. Lymph node involvement in the hilum region of the liver is eligible if the nodes do not exceed 2 cm.
* Known sensitivity to porphyrin-type drugs or known history of porphyria are exclusionary
* Pregnancy or breast-feeding patients are excluded. A negative pregnancy test (urine or serum) from women of childbearing age is required prior to enrollment. A fertile patient must use effective contraception during participation in the study
* Concurrent participation in another clinical trial involving experimental treatment is excluded
* Any concurrent disease or condition that in the opinion of the investigator impairs the patient's ability to complete the trial such as psychological, familial, sociological, geographical or medical conditions which in the Principal Investigator's opinion could compromise compliance with the objectives and procedures of this protocol or obscure interpretation of the trial's data are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2006-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 130 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sy-Shi Wang, PhD, Study Director — Light Sciences Oncology
Locations (34):
- University Hospital Dubrava, Zagreb, Croatia
- Hong Kong (2):
  - Tuen Mun Hospital, Tuenmen, New Territories
  - Prince of Wales Hospital, Dept. of Clincal Oncology, New Territories
- India (5):
  - Dr. Kamakshi Memorial Hospital, Chennai
  - SMS Medical College, Jaipur
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - Cancer Clinic, Nagpur
  - Shatabdi Super Specialty Hospital, Nashik
- Malaysia (4):
  - Island Hospital, George Town
  - Lam Wah Ee Hospital, George Town
  - Hospital Universiti Kebangsaan Malaysia, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Philippines (6):
  - Cebu Doctors University Hospital, Cebu City
  - Vicente Sotto Memorial Medical Center, Cebu City
  - Santo Tomas University Hospital, Manila
  - The Medical City, Pasig
  - National Kidney and Transplant Institute, Quezon City
  - St. Luke's Medical Center, Quezon City
- Poland (2):
  - Szpital Uniwersytecki CMUJ, Krakow
  - Centralny Szpital Kliniczny MSWiA, Warsaw
- Serbia (3):
  - Clinical Center of Serbia, Institute for Gastroenterology and Hepatology, Belgrade
  - Clinical Center of Serbia, Belgrade
  - Military Medical Academy, Belgrade
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Korea University Medical Center Anam Hospital, Seoul
  - Kyunghee Univeristy Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Sinchon Severance Hospital, Yonsei University, Seoul
- Karolinska University Hospital, Stockholm, Sweden
- Thailand (2):
  - Mahidol University, Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai